CLINICAL TRIAL: NCT01994889
Title: A MULTICENTER, INTERNATIONAL, PHASE 3, DOUBLE-BLIND, PLACEBO-CONTROLLED, RANDOMIZED STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF DAILY ORAL DOSING OF TAFAMIDIS MEGLUMINE (PF-06291826) 20 MG OR 80 MG IN COMPARISON TO PLACEBO IN SUBJECTS DIAGNOSED WITH TRANSTHYRETIN CARDIOMYOPATHY (TTR-CM)
Brief Title: Safety and Efficacy of Tafamidis in Patients With Transthyretin Cardiomyopathy
Acronym: ATTR-ACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3461028; 2012-002465-35 (EudraCT Number); ATTR-ACT (Other: Alias Study Number)
Record Dates: First submitted 2013-11-14; First posted 2013-11-26 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Transthyretin (TTR) Amyloid Cardiomyopathy
Keywords: amyloidosis; amyloid; transthyretin; TTR
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Alzheimer Disease | interventions — tafamidis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tafamidis - 20 mg (Experimental): Active Treatment-Low dose
  Interventions: Drug: Tafamidis
- Tafamidis - 80 mg (Experimental): Active Treatment-High Dose
  Interventions: Drug: Tafamidis
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafamidis — Tafamidis 20 mg in soft gel capsules administered once a day for 30 months
  Arms: Tafamidis - 20 mg
Drug: Tafamidis — Tafamidis 80 mg in soft gel capsules administered once a day for 30 months
  Arms: Tafamidis - 80 mg
Drug: Placebo — Placebo in soft gel capsules administered once a day for 30 months
  Arms: Placebo

SUMMARY:
This Phase 3 study will investigate the efficacy, safety and tolerability of an oral daily dose of 20 mg or 80 mg tafamidis meglumine capsules compared to placebo in subjects with either transthyretin genetic variants or wild-type transthyretin resulting in amyloid cardiomyopathy.

DETAILED DESCRIPTION:
Phase 3, multicenter, global, three-arm, parallel design, placebo-controlled, double-blind, randomized study to determine efficacy, safety and tolerability of tafamidis on clinical outcomes (all-cause mortality and frequency of cardiovascular-related hospitalizations) in subjects with either transthyretin genetic variants or wild-type transthyretin resulting in amyloid cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of Heart Failure (HF) with at least 1 prior hospitalization for HF or clinical evidence of HF (without hospitalization) manifested by signs or symptoms of volume overload or elevated intracardiac pressures (e.g., elevated jugular venous pressure, shortness of breath or signs of pulmonary congestion on x-ray or auscultation, peripheral edema) that required/requires treatment with a diuretic for improvement,
* Evidence of cardiac involvement by echocardiography with an end-diastolic interventricular septal wall thickness > 12 mm,
* Presence of amyloid deposits in biopsy tissue and presence of a variant TTR genotype and/or TTR precursor protein identification by immunohistochemistry, scintigraphy or mass spectrometry

Exclusion Criteria:

* A New York Heart Association (NYHA) classification of IV.
* Presence of primary (light chain) amyloidosis.
* Prior liver or heart transplantation or implanted cardiac mechanical assist device.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- United States (50):
  - The Kirklin Clinic, Birmingham, Alabama
  - UAB Hospital Department of Pharmacy IDS, Birmingham, Alabama
  - University Hospital, University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona - Mayo Clinic Speciality Building, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona - Mayo Clinic Building, Scottsdale, Arizona
  - UCSD Clinical and Translational Research Institute, Investigational Drug Service, La Jolla, California
  - Altman Clinical Translational Research institute, La Jolla, California
  - Altman Clinical Translational Research Institute, La Jolla, California
  - UCSD Sulpizio Cardiovascular Center, La Jolla, California
  - Cedars-Sinai Medical Center, Investigational Drug Pharmacy Services, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Care Foundation, Los Angeles, California
  - UCSF Cardiovascular Care and Prevention Center, San Francisco, California
  - Stanford University Hospital and Clinics, Stanford, California
  - UM Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Christ Medical Centre, Oak Lawn, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - The Johns Hopkins Hospital IDS Pharmacy, Baltimore, Maryland
  - Boston Medical Center - Cardiovascular Center, Outpatient Clinic, Boston, Massachusetts
  - Boston Medical Center Investigational Pharmacy Services, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston University Medical Center General Clinical Research Unit, Boston, Massachusetts
  - Michigan Medicine,University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Pharmacy Research Supp, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York University Hospitals, New York, New York
  - Icahn School of Medicine at Mount Sinai and Mount Sinai Hospital, New York, New York
  - Mount Sinai Doctors Faculty Practice, New York, New York
  - The Mount Sinai Hospital Department of Pharmacy, New York, New York
  - Columbia University Medical Center Research Pharmacy, New York, New York
  - Columbia University Medical Center/Clinical Cardiovascular Research Laboratory for the Elderly, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health and Science University (OHSU), Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah,Health Sciences Center, Salt Lake City, Utah
  - VCU Medical Center - Ambulatory Care Clinic, Richmond, Virginia
  - VCU Medical Center - Main Hospital, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Unidade de Pesquisa Clinica / Hospital Universitario Clementino Fraga Filho / UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (2):
  - University of Calgary/Foothills Medical Centre, Calgary, Alberta
  - Toronto General Hospital, Toronto, Ontario
- Czechia (6):
  - Fakultni nemocnice u sv. Anny, Nemocnicni lekarna, Brno
  - Nemocnice u sv. Anny v Brne, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Vseobecna fakultni nemocnice v Praze, Nemocnicni lekarna, Prague
  - IKEM, Ustavni lekarna, Prague
  - IKEM, Prague
- France (2):
  - Hopital Antoine Beclere, Clamart
  - CHU Henri Mondor, Créteil
- Germany (2):
  - Medical University of Heidelberg, Heidelberg
  - Universitaetsklinikum Muenster, Münster
- Italy (4):
  - U.O. Cardiologia- Prof. Rapezzi, Bologna
  - Unita Operativa di Cardiologia, Brescia
  - S.O.D. Cardiologia Generale 1 - D.A.I. del Cuore e dei Vasi, Florence
  - Centro per lo Studio e la Cura Delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico S. Matteo, Pavia
- Japan (3):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shinshu University Hospital, Nagano
- University Medical Center Groningen, Groningen, Netherlands
- Spain (3):
  - Hospital Universitario Puerta De Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario A Coruna, A Coruña
- Sweden (2):
  - Medicin-Geriatrik kliniken-Skelleftea lasarett, Skellefteå
  - Sjukhusvägen, Akademiska sjukhuset, Uppsala
- United Kingdom (3):
  - St Bartholomew's Hospital-Barts Health NHS Trust, London
  - St. George's Hospital (St George's Healthcare NHS Trust), London
  - St. George's University of London, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Damy T, Wang R, Maurer MS, Gillmore JD, Fontana M. Long-term efficacy of tafamidis in patients with transthyretin amyloid cardiomyopathy by National Amyloidosis Centre stage. Eur J Heart Fail. 2025 Jun 9. doi: 10.1002/ejhf.3696. Online ahead of print. PMID 40488446
- [Derived] Grogan M, Davis MK, Crespo Leiro MG, Sultan MB, Gundapaneni B, Angeli FS, Hanna M. The effect of long-term tafamidis treatment on quality of life in people with transthyretin amyloid cardiomyopathy (ATTR-CM): A plain language summary. Future Cardiol. 2024;20(11-12):595-603. doi: 10.1080/14796678.2024.2391250. Epub 2024 Sep 11. PMID 39258729
- [Derived] Witteles R, Jefferies JL, Kapa S, Cappelli F, Sultan MB, Gundapaneni B, Davis MK, Garcia-Pavia P. Atrial Fibrillation as a Prognostic Factor for All-Cause Mortality in Patients With Transthyretin Amyloid Cardiomyopathy. JACC CardioOncol. 2024 Apr 30;6(4):592-598. doi: 10.1016/j.jaccao.2024.03.007. eCollection 2024 Aug. PMID 39239341
- [Derived] Hanna M, Fine NM, Gundapaneni B, Sultan MB, Witteles RM. Improvements in Efficacy Measures With Tafamidis in the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial. JACC Adv. 2022 Dec 14;1(5):100148. doi: 10.1016/j.jacadv.2022.100148. eCollection 2022 Dec. PMID 38939456
- [Derived] Drachman B, Damy T, Hanna M, Wang R, Angeli FS, Garcia-Pavia P. Long-term tafamidis efficacy in patients with transthyretin amyloid cardiomyopathy by baseline left ventricular ejection fraction. Eur J Heart Fail. 2024 Sep;26(9):2038-2046. doi: 10.1002/ejhf.3330. Epub 2024 Jun 26. PMID 38932583
- [Derived] Sperry BW, Sultan MB, Gundapaneni B, Tai SS, Witteles RM. Effect of Tafamidis on Renal Function in Patients With Transthyretin Amyloid Cardiomyopathy in ATTR-ACT. JACC CardioOncol. 2024 Apr 16;6(2):300-306. doi: 10.1016/j.jaccao.2024.02.007. eCollection 2024 Apr. PMID 38774010
- [Derived] Shah SJ, Fine N, Garcia-Pavia P, Klein AL, Fernandes F, Weissman NJ, Maurer MS, Boman K, Gundapaneni B, Sultan MB, Elliott P. Effect of Tafamidis on Cardiac Function in Patients With Transthyretin Amyloid Cardiomyopathy: A Post Hoc Analysis of the ATTR-ACT Randomized Clinical Trial. JAMA Cardiol. 2024 Jan 1;9(1):25-34. doi: 10.1001/jamacardio.2023.4147. PMID 37966817
- [Derived] Garcia-Pavia P, Sultan MB, Gundapaneni B, Sekijima Y, Perfetto F, Hanna M, Witteles R. Tafamidis Efficacy Among Octogenarian Patients in the Phase 3 ATTR-ACT and Ongoing Long-Term Extension Study. JACC Heart Fail. 2024 Jan;12(1):150-160. doi: 10.1016/j.jchf.2023.08.032. Epub 2023 Nov 8. PMID 37943223
- [Derived] Elliott P, Gundapaneni B, Sultan MB, Ines M, Garcia-Pavia P. Improved long-term survival with tafamidis treatment in patients with transthyretin amyloid cardiomyopathy and severe heart failure symptoms. Eur J Heart Fail. 2023 Nov;25(11):2060-2064. doi: 10.1002/ejhf.2974. Epub 2023 Jul 26. PMID 37434378
- [Derived] Bhambri R, Colavecchia AC, Bruno M, Chen Y, Alvir J, Roy A, Kemner J, Crowley A, Benjumea D, Gilstrap L. Real-World Characteristics of Patients with Wild-Type Transthyretin Amyloid Cardiomyopathy: An Analysis of Electronic Healthcare Records in the United States. Am J Cardiovasc Drugs. 2023 Mar;23(2):197-206. doi: 10.1007/s40256-022-00563-4. Epub 2023 Feb 13. PMID 36780092
- [Derived] Sperry BW, Hanna M, Maurer MS, Nativi-Nicolau J, Floden L, Stewart M, Wyrwich KW, Barsdorf AI, Kapadia H, Spertus JA. Association of Tafamidis With Health Status in Patients With ATTR Cardiac Amyloidosis: A Post Hoc Analysis of the ATTR-ACT Randomized Clinical Trial. JAMA Cardiol. 2023 Mar 1;8(3):275-280. doi: 10.1001/jamacardio.2022.5251. PMID 36723935
- [Derived] Elliott P, Drachman BM, Gottlieb SS, Hoffman JE, Hummel SL, Lenihan DJ, Ebede B, Gundapaneni B, Li B, Sultan MB, Shah SJ. Long-term survival in people with transthyretin amyloid cardiomyopathy who took tafamidis: A Plain Language Summary. Future Cardiol. 2023 Jan;19(1):7-17. doi: 10.2217/fca-2022-0096. Epub 2023 Jan 30. PMID 36715498
- [Derived] Tess DA, Maurer TS, Li Z, Bulawa C, Fleming J, Moody AT. Relationship of binding-site occupancy, transthyretin stabilisation and disease modification in patients with tafamidis-treated transthyretin amyloid cardiomyopathy. Amyloid. 2023 Jun;30(2):208-219. doi: 10.1080/13506129.2022.2145876. Epub 2022 Nov 18. PMID 36399070
- [Derived] Maeda-Ogata S, Tahara N, Tahara A, Bekki M, Honda A, Sugiyama Y, Igata S, Abe T, Sekijima Y, Ueda M, Ando Y, Fukumoto Y. Treatment response to Tafamidis quantitatively assessed by serial bone scintigraphy in transthyretin amyloid cardiomyopathy. J Nucl Cardiol. 2023 Feb;30(1):403-404. doi: 10.1007/s12350-022-03137-8. Epub 2022 Nov 8. No abstract available. PMID 36348245
- [Derived] Rozenbaum MH, Tran D, Bhambri R, Nativi-Nicolau J. Annual Cardiovascular-Related Hospitalization Days Avoided with Tafamidis in Patients with Transthyretin Amyloid Cardiomyopathy. Am J Cardiovasc Drugs. 2022 Jul;22(4):445-450. doi: 10.1007/s40256-022-00526-9. Epub 2022 Mar 30. PMID 35353352
- [Derived] Nativi-Nicolau J, Judge DP, Hoffman JE, Gundapaneni B, Keohane D, Sultan MB, Grogan M. How did transthyretin amyloid cardiomyopathy progress in patients who took placebo in the study ATTR-ACT? A plain language summary. Future Cardiol. 2022 Mar 17. doi: 10.2217/fca-2021-0150. Online ahead of print. PMID 35297655
- [Derived] Elliott P, Drachman BM, Gottlieb SS, Hoffman JE, Hummel SL, Lenihan DJ, Ebede B, Gundapaneni B, Li B, Sultan MB, Shah SJ. Long-Term Survival With Tafamidis in Patients With Transthyretin Amyloid Cardiomyopathy. Circ Heart Fail. 2022 Jan;15(1):e008193. doi: 10.1161/CIRCHEARTFAILURE.120.008193. Epub 2021 Dec 20. PMID 34923848
- [Derived] Hanna M, Damy T, Grogan M, Stewart M, Gundapaneni B, Sultan MB, Maurer MS. Tafamidis and quality of life in people with transthyretin amyloid cardiomyopathy in the study ATTR-ACT: A plain language summary. Future Cardiol. 2022 Mar;18(3):165-172. doi: 10.2217/fca-2021-0095. Epub 2021 Nov 15. PMID 34779246
- [Derived] Rozenbaum MH, Garcia A, Grima D, Tran D, Bhambri R, Stewart M, Li B, Heeg B, Postma M, Masri A. Health impact of tafamidis in transthyretin amyloid cardiomyopathy patients: an analysis from the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial (ATTR-ACT) and the open-label long-term extension studies. Eur Heart J Qual Care Clin Outcomes. 2022 Aug 17;8(5):529-538. doi: 10.1093/ehjqcco/qcab031. PMID 33895806
- [Derived] Vong C, Boucher M, Riley S, Harnisch LO. Modeling of Survival and Frequency of Cardiovascular-Related Hospitalization in Patients with Transthyretin Amyloid Cardiomyopathy Treated with Tafamidis. Am J Cardiovasc Drugs. 2021 Sep;21(5):535-543. doi: 10.1007/s40256-021-00464-y. Epub 2021 Mar 26. PMID 33770392
- [Derived] Miller AB, Januzzi JL, O'Neill BJ, Gundapaneni B, Patterson TA, Sultan MB, Lopez-Sendon J. Causes of Cardiovascular Hospitalization and Death in Patients With Transthyretin Amyloid Cardiomyopathy (from the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial [ATTR-ACT]). Am J Cardiol. 2021 Jun 1;148:146-150. doi: 10.1016/j.amjcard.2021.02.035. Epub 2021 Mar 3. PMID 33667442
- [Derived] Rapezzi C, Elliott P, Damy T, Nativi-Nicolau J, Berk JL, Velazquez EJ, Boman K, Gundapaneni B, Patterson TA, Schwartz JH, Sultan MB, Maurer MS. Efficacy of Tafamidis in Patients With Hereditary and Wild-Type Transthyretin Amyloid Cardiomyopathy: Further Analyses From ATTR-ACT. JACC Heart Fail. 2021 Feb;9(2):115-123. doi: 10.1016/j.jchf.2020.09.011. Epub 2020 Dec 9. PMID 33309574
- [Derived] Hanna M, Damy T, Grogan M, Stewart M, Gundapaneni B, Patterson TA, Schwartz JH, Sultan MB, Maurer MS. Impact of Tafamidis on Health-Related Quality of Life in Patients With Transthyretin Amyloid Cardiomyopathy (from the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial). Am J Cardiol. 2021 Feb 15;141:98-105. doi: 10.1016/j.amjcard.2020.10.066. Epub 2020 Nov 19. PMID 33220323
- [Derived] Damy T, Garcia-Pavia P, Hanna M, Judge DP, Merlini G, Gundapaneni B, Patterson TA, Riley S, Schwartz JH, Sultan MB, Witteles R. Efficacy and safety of tafamidis doses in the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial (ATTR-ACT) and long-term extension study. Eur J Heart Fail. 2021 Feb;23(2):277-285. doi: 10.1002/ejhf.2027. Epub 2020 Nov 12. PMID 33070419
- [Derived] Li B, Alvir J, Stewart M. Extrapolation of Survival Benefits in Patients with Transthyretin Amyloid Cardiomyopathy Receiving Tafamidis: Analysis of the Tafamidis in Transthyretin Cardiomyopathy Clinical Trial. Cardiol Ther. 2020 Dec;9(2):535-540. doi: 10.1007/s40119-020-00179-2. Epub 2020 Jun 10. PMID 32524297
- [Derived] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Derived] Maurer MS, Elliott P, Merlini G, Shah SJ, Cruz MW, Flynn A, Gundapaneni B, Hahn C, Riley S, Schwartz J, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Design and Rationale of the Phase 3 ATTR-ACT Clinical Trial (Tafamidis in Transthyretin Cardiomyopathy Clinical Trial). Circ Heart Fail. 2017 Jun;10(6):e003815. doi: 10.1161/CIRCHEARTFAILURE.116.003815. PMID 28611125
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461028&StudyName=Safety%20and%20Efficacy%20of%20Tafamidis%20in%20Patients%20with%20Transthyretin%20Cardiomyopathy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pooled analysis of the tafamidis treatment groups [20 milligrams (mg) and 80 mg] was performed in comparison to placebo group.
Groups:
- Tafamidis 20 mg: Participants with variant transthyretin cardiomyopathy (TTR-CM) genotype or wild-type TTR-CM genotype received one tafamidis 20 milligram (mg) capsule + 3 placebo capsules (matched to tafamidis) orally once daily for 30 months.
- Tafamidis 80 mg: Participants with variant TTR-CM genotype or wild-type TTR-CM genotype received tafamidis 80 mg (4 capsules of 20 mg each) orally once daily for 30 months.
- Placebo: Participants with variant TTR-CM genotype or wild-type TTR-CM genotype received 4 placebo capsules matched to tafamidis orally once daily for 30 months.
Period: Overall Study
Arm/Group | Tafamidis 20 mg | Tafamidis 80 mg | Placebo
Started | 88 | 176 | 177
Completed | 60 | 113 | 85
Not Completed | 28 | 63 | 92
Not completed — Adverse Event | 5 | 12 | 11
Not completed — Cardiac Device Implantation | 0 | 2 | 0
Not completed — Organ Transplantation | 1 | 5 | 5
Not completed — No longer willing to participate | 8 | 17 | 37
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Death | 14 | 25 | 38

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all participants in the safety population (all randomized participants who received at least 1 dose of double-blind medication) who had at least 1 post baseline efficacy evaluation ( post baseline hospitalization, study visit, or date of death).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafamidis 20 mg | Tafamidis 80 mg | Placebo | Total
Number analyzed (Participants) | 88 | 176 | 177 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (7.07) | 75.2 (7.24) | 74.1 (6.69) | 74.3 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 18 | 20 | 43
  Male | 83 | 158 | 157 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7 | 14
  Not Hispanic or Latino | 84 | 171 | 170 | 425
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 11 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 26 | 26 | 63
  White | 75 | 136 | 146 | 357
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Combination of All-Cause Mortality and Frequency of Cardiovascular-Related Hospitalizations
Description: All-cause mortality and frequency of cardiovascular hospitalization were analyzed using Finkelstein-Schoenfeld method. The method combines all-cause mortality and frequency of CV-related hospitalizations in a hierarchical fashion using all-cause mortality first. The method compares every participant with every other participant within strata, assigning a +1 to the "better" participant and a -1 to the "worse" participant and 0 if they are "tied". Participants who discontinued for transplantation (heart transplantation and combined heart and liver transplantation) or for implantation of a cardiac mechanical assist device, were handled in the same manner as death. 'Win' represents a participant doing better based on hierarchical comparison. The reported unit is the total "wins" for each treatment group from performing such a hierarchical comparison across all 4 strata in the study.
Time Frame: Baseline up to Month 30
Population: ITT analysis set:participants in safety population(randomized participants who received at least 1 dose of double-blind medication)having at least 1 post baseline efficacy.Pre-specified intent of study was to compare results between tafamidis with placebo,irrespective of tafamidis doses. Analysis based on pooled dose groups,as per study protocol.
Measure: Number; unit: wins
Groups:
- Tafamidis: Participants with variant TTR-CM genotype or wild-type TTR-CM genotype received one tafamidis 20 mg + 3 placebo capsules (matched to tafamidis) or 80 mg (4 capsules of 20 mg each) capsule orally once daily for 30 months.
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
wins | 8595 | 5071
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Test type: Superiority; p = 0.0006, Finkelstein-Schoenfeld Method

2. Secondary Outcome: All-Cause Mortality
Description: Number of deaths due to any cause was analyzed. Participants who discontinued for transplantation (heart transplantation and combined heart and liver transplantation) or for implantation of a cardiac mechanical assist device were handled in the same manner as death.
Time Frame: Baseline up to Month 30
Population: ITT analysis set: all participants in the safety population who had at least 1 post baseline efficacy evaluation. The pre-specified intent of this study was to compare the results between tafamidis with placebo, irrespective of the tafamidis doses. Therefore, this analysis was based on the pooled dose groups, as per the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
Participants
  Deaths (all causes) | 69 | 72
  Heart transplants | 7 | 4
  Cardiac Mechanical Assist Devices | 2 | 0
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Test type: Superiority; p = 0.0259, Cox proportional hazards model; Hazard Ratio (HR) = 0.698, 95% CI 2-sided [0.508 to 0.958] — Hazard ratio from a Cox proportional hazards model with treatment, TTR genotype (variant and wild-type) and New York Heart Association (NYHA) baseline classification (NYHA Classes I and II combined and NYHA Class III) in the model

3. Secondary Outcome: Frequency of Cardiovascular-Related Hospitalizations
Description: CV related hospitalizations per year is calculated as participant's number of CV related hospitalizations upon duration on study in years.
Time Frame: Baseline to Month 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: CV hospitalization per year
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
CV hospitalization per year | 0.999 (2.2777) | 0.884 (1.2032)
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Test type: Superiority; p < 0.0001, Poisson regression analysis — Poisson regression analysis with treatment, TTR genotype, NYHA baseline classification, treatment-by-TTR genotype interaction, and treatment-by-NYHA baseline classification interaction terms as factors adjusted for treatment duration; Risk Ratio (RR) = 0.6761, 95% CI 2-sided [0.5639 to 0.8107]

4. Secondary Outcome: Change From Baseline in the Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 30
Description: 6MWT is the total distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Baseline, Month 30
Population: Analysis performed on ITT analysis set. The pre-specified intent of this study was to compare the results between tafamidis with placebo, irrespective of the tafamidis doses. This analysis was based on the pooled dose groups, as per the study protocol. Here, 'number analyzed' = participants evaluable for this outcome at specified time points.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
meters
  Baseline | 350.55 (121.296) | 353.26 (125.983)
  Change at Month 30: number analyzed (Participants) | 155 | 70
  Change at Month 30 | -30.46 (87.886) | -89.67 (105.159)
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; L.S. means are from an ANCOVA (MMRM) model with an unstructured covariance matrix; center and participant within center as random effects; treatment, visit, TTR genotype (variant and wild-type), and visit by treatment interaction, as fixed effects and baseline score as covariate; Test type: Superiority; p < .0001, Mixed Model Repeated Measures ANCOVA; Least Square Mean Difference = 75.68, 95% CI 2-sided [57.56 to 93.80], Standard Error of Mean 9.236

5. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) at Month 30
Description: KCCQ is a 23-item participant-completed questionnaire that assesses health status and health-related quality of life in participants with heart failure. Eight domain scores were calculated for the KCCQ: Physical limitation, Social limitation, Quality of life, Self-efficacy, Symptom stability, Symptom frequency, Symptom burden, and Total symptoms (calculated as the mean of Symptom frequency and Symptom burden scores). Two summary scores were also calculated: Clinical Summary (calculated as mean of Physical limitation and Total symptom scores) and Overall Summary (calculated as mean of Physical limitation, Social limitation, Total symptoms, and Quality of life scores). Domain and summary scores were scaled to range from 0 (minimum) to 100 (maximum); higher scores represent better health status.
Time Frame: Baseline, Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
units on a scale
  Baseline | 67.274 (21.3561) | 65.898 (21.7357)
  Change at Month 30: number analyzed (Participants) | 170 | 84
  Change at Month 30 | -3.855 (19.3075) | -14.637 (21.4078)
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Change at Month 30; Test type: Superiority; p < .0001, Mixed Model Repeated Measures ANCOVA; LS Mean Difference = 13.65, 95% CI 2-sided [9.48 to 17.83], Standard Error of Mean 2.130

6. Secondary Outcome: Number of Participants With Cardiovascular-Related Mortality
Description: Deaths adjudicated as CV-related and indeterminate are reported. Participants who discontinued for transplantation (heart transplantation and combined heart and liver transplantation) or for implantation of a cardiac mechanical assist device, were handled in the same manner as death.
Time Frame: Baseline up to Month 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 264 | 177
Participants | 64 | 63
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Test type: Superiority; p = 0.0383, Cox proportional hazards model; Hazard Ratio (HR) = 0.691, 95% CI 2-sided [0.488 to 0.980] — Hazard ratio from a Cox proportional hazards model with treatment, TTR genotype (variant and wild-type) and NYHA baseline classification (NYHA Classes I and II combined and NYHA Class III) in the model

7. Secondary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR) at Month 1
Description: TTR stabilization is a measure of the degree of stabilization afforded the TTR molecule by tafamidis.
Time Frame: Month 1
Population: Analysis performed on ITT analysis set. The pre-specified intent of this study was to compare the results between tafamidis with placebo, irrespective of the tafamidis doses. This analysis was based on the pooled dose groups, as per the study protocol. Here, 'number of participants analyzed' = participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Tafamidis | Placebo
Number analyzed (Participants) | 245 | 170
percentage of participants | 86.1 | 3.5
Statistical Analysis 1: Comparison: Tafamidis vs Placebo; Test type: Superiority; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (Month 31)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Tafamidis 20 mg | Tafamidis 80 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 23/88 | 49/176 | 72/177
Serious Adverse Events (participants affected / at risk) | 66/88 | 133/176 | 140/177
Other Adverse Events (participants affected / at risk) | 86/88 | 170/176 | 171/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=88) | Tafamidis 80 mg (N=176) | Placebo (N=177)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 3
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 11 | 8
Atrial flutter (Cardiac disorders) | 2 | 4 | 5
Atrial tachycardia (Cardiac disorders) | 1 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 4 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 5 | 5
Cardiac amyloidosis (Cardiac disorders) | 2 | 3 | 5
Cardiac arrest (Cardiac disorders) | 1 | 2 | 6
Cardiac failure (Cardiac disorders) | 16 | 34 | 39
Cardiac failure acute (Cardiac disorders) | 4 | 23 | 17
Cardiac failure chronic (Cardiac disorders) | 1 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 15 | 20 | 32
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 3 | 2 | 4
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2
Left ventricular failure (Cardiac disorders) | 1 | 3 | 6
Myocardial depression (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 2
Systolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 3
Ventricular tachycardia (Cardiac disorders) | 2 | 2 | 7
Familial amyloidosis (Congenital, familial and genetic disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 3 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 2 | 4 | 2
Disease progression (General disorders) | 1 | 4 | 3
General physical health deterioration (General disorders) | 1 | 0 | 2
Generalised oedema (General disorders) | 1 | 0 | 1
Incarcerated hernia (General disorders) | 0 | 0 | 1
Medical device site haematoma (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 4 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Amyloidosis (Immune system disorders) | 1 | 1 | 2
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Necrotising soft tissue infection (Infections and infestations) | 0 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 13 | 12
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 1 | 2
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 1 | 1
Serratia infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 5
Urosepsis (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 9 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 1 | 1
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 2 | 6
Fluid retention (Metabolism and nutrition disorders) | 2 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 4
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 5
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 6 | 10
Transient ischaemic attack (Nervous system disorders) | 3 | 1 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Device connection issue (Product Issues) | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 1
Device malfunction (Product Issues) | 0 | 2 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 4
Stress (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 13 | 15
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2 | 3
Renal impairment (Renal and urinary disorders) | 1 | 1 | 1
Renal injury (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=88) | Tafamidis 80 mg (N=176) | Placebo (N=177)
Anaemia (Blood and lymphatic system disorders) | 5 | 10 | 13
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 1
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6 | 5
Accelerated idioventricular rhythm (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 3 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 5 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 2 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 13 | 28 | 31
Atrial flutter (Cardiac disorders) | 5 | 8 | 12
Atrial tachycardia (Cardiac disorders) | 3 | 6 | 7
Atrial thrombosis (Cardiac disorders) | 1 | 1 | 4
Atrioventricular block (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 2 | 3
Atrioventricular block first degree (Cardiac disorders) | 2 | 3 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 2 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 3
Bundle branch block right (Cardiac disorders) | 0 | 1 | 2
Cardiac amyloidosis (Cardiac disorders) | 0 | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 18 | 20 | 33
Cardiac failure acute (Cardiac disorders) | 0 | 3 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 3 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 3
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Hepatojugular reflux (Cardiac disorders) | 2 | 3 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 2
Low cardiac output syndrome (Cardiac disorders) | 0 | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 2 | 6
Palpitations (Cardiac disorders) | 2 | 4 | 8
Pericardial effusion (Cardiac disorders) | 2 | 2 | 2
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 1
Rhythm idioventricular (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 3
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 6 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 2 | 4
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 3 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 5 | 6
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 3 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 5 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 2
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 3 | 2
Hypogonadism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 5 | 12 | 10
Thyroid mass (Endocrine disorders) | 1 | 1 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Blepharochalasis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 3 | 8 | 2
Chalazion (Eye disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 0
Diplopia (Eye disorders) | 2 | 0 | 2
Dry eye (Eye disorders) | 0 | 4 | 5
Eye disorder (Eye disorders) | 0 | 1 | 1
Eye haemorrhage (Eye disorders) | 0 | 1 | 2
Eye oedema (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Eyelid bleeding (Eye disorders) | 0 | 0 | 1
Eyelid cyst (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 1
Lacrimal structural disorder (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 0
Macular degeneration (Eye disorders) | 2 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1 | 0
Optic atrophy (Eye disorders) | 0 | 1 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 1 | 1 | 0
Scleral discolouration (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 2 | 5 | 3
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 2 | 3 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 6 | 7
Abdominal distension (Gastrointestinal disorders) | 6 | 7 | 5
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 8 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 5
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 7 | 6 | 9
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 14 | 25 | 30
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 22 | 39
Diverticulum (Gastrointestinal disorders) | 1 | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 5
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 4 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 8 | 3
Frequent bowel movements (Gastrointestinal disorders) | 0 | 3 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 1 | 3
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 0 | 7
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 4 | 4
Hiatus hernia (Gastrointestinal disorders) | 1 | 2 | 2
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 5 | 5 | 3
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 20 | 36
Oesophageal mass (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 2
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 2
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6 | 16
Asthenia (General disorders) | 11 | 16 | 11
Atrophy (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 3 | 8 | 8
Chest pain (General disorders) | 3 | 7 | 8
Chills (General disorders) | 2 | 2 | 2
Condition aggravated (General disorders) | 0 | 1 | 1
Cyst rupture (General disorders) | 0 | 1 | 0
Decreased activity (General disorders) | 0 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Early satiety (General disorders) | 2 | 2 | 3
Effusion (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 1 | 4
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 16 | 29 | 33
Feeling abnormal (General disorders) | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 4 | 4 | 11
General physical health deterioration (General disorders) | 1 | 4 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 1 | 1 | 2
Implant site haematoma (General disorders) | 2 | 0 | 1
Implant site pain (General disorders) | 2 | 1 | 1
Inflammation (General disorders) | 0 | 3 | 1
Influenza like illness (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 2 | 4
Mass (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 7 | 11 | 20
Oedema peripheral (General disorders) | 17 | 29 | 31
Pain (General disorders) | 1 | 6 | 2
Peripheral swelling (General disorders) | 2 | 6 | 7
Pseudocyst (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 4
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Temperature intolerance (General disorders) | 1 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 0 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 2 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 2 | 4 | 2
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 3 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Dust allergy (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 2 | 2
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bacterial abdominal infection (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 1
Body tinea (Infections and infestations) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 7 | 21 | 19
Candida infection (Infections and infestations) | 0 | 2 | 0
Candiduria (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 6 | 6 | 10
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 2
Cystitis (Infections and infestations) | 2 | 5 | 0
Device related infection (Infections and infestations) | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 2 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 2 | 0
Eye infection (Infections and infestations) | 0 | 2 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 2 | 0 | 2
Gas gangrene (Infections and infestations) | 0 | 0 | 1
Gastritis viral (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 5 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 3
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0 | 3
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 6 | 6
Hordeolum (Infections and infestations) | 0 | 2 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 4 | 7 | 6
Kidney infection (Infections and infestations) | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 2
Localised infection (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Lung infection (Infections and infestations) | 1 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 14 | 17
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 12 | 7
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 2 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 1 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 10 | 1
Skin infection (Infections and infestations) | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 17 | 16
Urinary tract infection (Infections and infestations) | 7 | 15 | 25
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Wound infection (Infections and infestations) | 0 | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bursa injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 11 | 5
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 24 | 38 | 40
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 5 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 3 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 6 | 3
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 4
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Metal poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 2
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Rib fracture (Injury, poisoning and procedural complications) | 2 | 2 | 3
Scar (Injury, poisoning and procedural complications) | 0 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 5 | 5
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 4 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 4
Anticoagulation drug level below therapeutic (Investigations) | 1 | 1 | 0
Arterial bruit (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1
Bence Jones protein urine present (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 3 | 1
Blood chloride decreased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Blood creatinine abnormal (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 9 | 8
Blood glucose increased (Investigations) | 0 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 1
Blood potassium abnormal (Investigations) | 0 | 0 | 2
Blood potassium decreased (Investigations) | 1 | 4 | 5
Blood potassium increased (Investigations) | 0 | 0 | 4
Blood pressure decreased (Investigations) | 0 | 0 | 2
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood pressure systolic decreased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 5
Blood urea increased (Investigations) | 3 | 8 | 5
Blood uric acid increased (Investigations) | 3 | 8 | 5
Blood urine present (Investigations) | 0 | 2 | 0
Body temperature decreased (Investigations) | 0 | 2 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 3
C-reactive protein increased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 2 | 3 | 4
Crystal urine present (Investigations) | 0 | 1 | 0
Drug level above therapeutic (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 5
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 9 | 11
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Heart rate decreased (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 2
Heart rate irregular (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Human epidermal growth factor receptor decreased (Investigations) | 0 | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 1 | 0
Inflammatory marker increased (Investigations) | 1 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 5 | 4 | 4
Liver function test abnormal (Investigations) | 0 | 0 | 2
Liver function test increased (Investigations) | 2 | 5 | 2
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 2 | 1
Occult blood positive (Investigations) | 0 | 0 | 2
Optic nerve cup/disc ratio increased (Investigations) | 1 | 0 | 0
Oxygen saturation abnormal (Investigations) | 0 | 2 | 2
Oxygen saturation decreased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 1 | 2
Prostatic specific antigen increased (Investigations) | 0 | 0 | 2
Protein urine present (Investigations) | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 3 | 3 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 1
Pulse absent (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Thyroid function test abnormal (Investigations) | 0 | 0 | 1
Thyroxine decreased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 2 | 3
Troponin increased (Investigations) | 1 | 2 | 4
Urobilinogen urine increased (Investigations) | 0 | 1 | 0
Venous pressure jugular abnormal (Investigations) | 0 | 0 | 1
Venous pressure jugular increased (Investigations) | 4 | 4 | 9
Vitamin D decreased (Investigations) | 0 | 2 | 2
Waist circumference increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 6 | 8 | 18
Weight increased (Investigations) | 7 | 13 | 12
White blood cell count decreased (Investigations) | 0 | 1 | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 3 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 8 | 14 | 25
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 11 | 18 | 27
Fluid retention (Metabolism and nutrition disorders) | 3 | 5 | 15
Gout (Metabolism and nutrition disorders) | 10 | 17 | 29
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 8 | 10
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 9 | 7
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 14 | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 8 | 10
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 3
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Protein deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 17 | 20
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 17 | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 15 | 14
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 13 | 11
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 9 | 6
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 27 | 20
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Ageusia (Nervous system disorders) | 0 | 2 | 3
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 2 | 4 | 3
Anosmia (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0
Asterixis (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 2 | 15 | 2
Brain injury (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 2 | 2 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 5 | 4 | 4
Cognitive disorder (Nervous system disorders) | 0 | 0 | 3
Dementia (Nervous system disorders) | 2 | 1 | 4
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 16 | 25 | 32
Dizziness postural (Nervous system disorders) | 0 | 4 | 7
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 3 | 4
Encephalopathy (Nervous system disorders) | 0 | 2 | 2
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 9 | 11
Hemiparesis (Nervous system disorders) | 1 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 5 | 4 | 6
Hypotonia (Nervous system disorders) | 0 | 1 | 0
Incoherent (Nervous system disorders) | 0 | 1 | 0
Intention tremor (Nervous system disorders) | 3 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 3 | 3
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 0 | 2 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 4 | 5 | 4
Mental impairment (Nervous system disorders) | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neurodegenerative disorder (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 3 | 12
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 5 | 6
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 2 | 2
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 3 | 6
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 5
Sciatica (Nervous system disorders) | 0 | 1 | 3
Seizure (Nervous system disorders) | 0 | 1 | 0
Senile dementia (Nervous system disorders) | 1 | 0 | 0
Sensorimotor disorder (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 2 | 6
Syncope (Nervous system disorders) | 5 | 5 | 11
Tension headache (Nervous system disorders) | 1 | 0 | 0
Tinel's sign (Nervous system disorders) | 1 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 8
Tunnel vision (Nervous system disorders) | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0
Device computer issue (Product Issues) | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 2
Device inappropriate shock delivery (Product Issues) | 0 | 0 | 1
Device loosening (Product Issues) | 1 | 0 | 0
Device malfunction (Product Issues) | 0 | 1 | 0
Device stimulation issue (Product Issues) | 0 | 0 | 2
Acrophobia (Psychiatric disorders) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 8 | 5
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 3 | 4
Delirium (Psychiatric disorders) | 1 | 3 | 3
Depressed mood (Psychiatric disorders) | 0 | 0 | 3
Depression (Psychiatric disorders) | 6 | 7 | 8
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 12 | 20 | 22
Major depression (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 1
Organic brain syndrome (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Persecutory delusion (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 8 | 18
Azotaemia (Renal and urinary disorders) | 1 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 4 | 6 | 6
Dysuria (Renal and urinary disorders) | 2 | 1 | 2
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 10 | 8 | 15
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 3
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2 | 5
Renal cyst (Renal and urinary disorders) | 1 | 4 | 2
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 5 | 8 | 7
Renal impairment (Renal and urinary disorders) | 2 | 5 | 8
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 2
Renal mass (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 2 | 2
Urinary retention (Renal and urinary disorders) | 2 | 6 | 12
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 6 | 7
Breast engorgement (Reproductive system and breast disorders) | 0 | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 1 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 5 | 3
Cervix disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 | 3
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 4 | 9 | 6
Nipple pain (Reproductive system and breast disorders) | 1 | 1 | 3
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 20 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 27 | 51
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 13
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 14
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 31
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 5
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychomalacia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 12 | 15
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 6 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 4 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 7 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Immobile (Social circumstances) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 2
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 1
Bleeding varicose vein (Vascular disorders) | 1 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 2 | 6 | 8
Haemorrhage (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 3 | 4
Hypotension (Vascular disorders) | 11 | 19 | 17
Jugular vein distension (Vascular disorders) | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 8 | 5
Pallor (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 2
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Varicophlebitis (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 2 | 1 | 1
Haemorrhagic cyst (General disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 2
Gingivitis (Infections and infestations) | 1 | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT01994889/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT01994889/SAP_001.pdf